CLINICAL TRIAL: NCT03890666
Title: CONNected Electronic Inhalers Asthma Control Trial 1 ("CONNECT 1"), a 12-Week Treatment, Multicenter, Open-Label, Randomized, Parallel Group Comparison, Feasibility Study to Evaluate the Effectiveness of the Albuterol eMDPI Digital System, to Optimize Outcomes in Patients at Least 13 Years of Age or Older With Asthma
Brief Title: A 12-Week Treatment Study to Evaluate the Effectiveness of Albuterol Multidose Dry Powder Inhaler With Integrated Electronic Module Digital System (eMDPI DS) in Participants13 Years or Older With Asthma
Acronym: CONNECT1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABS-AS-40138
Record Dates: First submitted 2019-03-18; First posted 2019-03-26 (Actual); Results first posted 2022-10-27 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Digital System (DS) (Experimental): Participants will be trained on the use of the albuterol eMDPI DS (including instructions on how to use both the eMDPI and the App) and, upon demonstrating competency, will receive 2 albuterol eMDPI devices for use as reliever bronchodilators to replace their reliever treatment during the study. The eMDPI Digital System consists of 4 devices: Device 1: albuterol eMDPI (the test investigational medicinal product [IMP]); Device 2: Patient-facing App; Device 3: Digital health platform (DHP) (Cloud solution); and Device 4: Provider-facing Dashboard. Participants will receive 90 micrograms (mcg) albuterol, 1 to 2 oral inhalations every 4 to 6 hours, as needed for 12 weeks.
  Interventions: Drug: Albuterol eMDPI DS
- Concurrent Control (CC) (Active Comparator): Participants will be treated with their standard of care albuterol-administering reliever inhalers and will use the digital system during the treatment period. Participants will be reimbursed or given a voucher to use to purchase their existing reliever medications.
  Interventions: Drug: albuterol

INTERVENTIONS:
Drug: Albuterol eMDPI DS — Albuterol sulfate electronic multidose dry powder inhaler (Albuterol eMDPI) DS with 4 component devices:
  * Device 1: Albuterol eMDPI
  * Device 2: Albuterol eMDPI Patient-facing smart device application (App)
  * Device 3: DHP Cloud solution)
  * Device 4: Provider-facing dashboard (dashboard)
  Arms: Digital System (DS)
Drug: albuterol — Standard of care albuterol-administering rescue inhaler
  Arms: Concurrent Control (CC)

SUMMARY:
This is a 12-week treatment, multicenter, open-label, randomized, parallel group comparison feasibility study to evaluate the effectiveness of the Albuterol eMDPI Digital System (DS), including inhaler, App, digital health platform (DHP) (Cloud solution), and dashboard, to optimize outcomes in participants at least 13 years of age or older with asthma.

The study will consist of a screening visit, a 12-week open-label treatment period, and a follow-up telephone call (2 weeks following treatment completion).

Participants with suboptimal asthma control will be enrolled in the study and randomized in a 1:1 ratio to 1 of 2 parallel groups stratified by investigational center: DS group participants utilizing the Albuterol eMDPI DS, including inhaler, App, DHP (Cloud solution), and dashboard, and CC group participants who will be treated with their standard of care albuterol-administering rescue inhalers and will not use the DS during the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* The participant has a documented diagnosis of asthma
* The participant is currently on treatment with an inhaled corticosteroid (ICS) with a long-acting beta2 antagonist (LABA).
* The participant is currently using inhaled albuterol sulfate as rescue medication and is willing to discontinue all other rescue medications and replace them with the study provided Albuterol eMDPI.
* The participant can read and communicate in English and is familiar with and is willing to use his/her own smart device and download and use the App.

  * Additional criteria apply, please contact the investigator for more information

Exclusion Criteria:

* The participant has any clinically significant uncontrolled medical condition (treated or untreated) other than asthma.
* The participant was hospitalized for severe asthma in the last 30 days.
* The participant has a diagnosis of Chronic Obstructive Pulmonary Disease (COPD) or Asthma-COPD Overlap (ACO).
* The participant is a current smoker or has a greater than 10 pack-year history of smoking.
* The participant is currently being treated with systemic corticosteroids (oral, intramuscular, or intravenous) or has been treated within the last 30 days.
* The participant has any treatment with biologics for asthma (for example, omalizumab, anti-IL5, anti-IL5R, anti-IL4R), or has had such treatment within the last 90 days.

  * Additional criteria apply, please contact the investigator for more information

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2021-10-04 (Actual); Study Completion 2021-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (30):
- United States (30):
  - Teva Investigational Site 14232, Birmingham, Alabama
  - Teva Investigational Site 14302, Los Angeles, California
  - Teva Investigational Site 14301, Stockton, California
  - Teva Investigational Site 14236, Colorado Springs, Colorado
  - Teva Investigational Site 14198, Denver, Colorado
  - Teva Investigational Site 14220, New Haven, Connecticut
  - Teva Investigational Site 14197, Aventura, Florida
  - Teva Investigational Site 14306, Miami, Florida
  - Teva Investigational Site 14215, Sarasota, Florida
  - Teva Investigational Site 14304, Albany, Georgia
  - Teva Investigational Site 14201, Gainesville, Georgia
  - Teva Investigational Site 14195, Savannah, Georgia
  - Teva Investigational Site 14217, Evanston, Illinois
  - Teva Investigational Site 14218, Springfield, Illinois
  - Teva Investigational Site 14305, Louisville, Kentucky
  - Teva Investigational Site 14191, Owensboro, Kentucky
  - Teva Investigational Site 14233, Ann Arbor, Michigan
  - Teva Investigational Site 14207, Bellevue, Nebraska
  - Teva Investigational Site 14221, New York, New York
  - Teva Investigational Site 14234, Chapel Hill, North Carolina
  - Teva Investigational Site 14187, Cincinnati, Ohio
  - Teva Investigational Site 14210, Philadelphia, Pennsylvania
  - Teva Investigational Site 14208, Pittsburgh, Pennsylvania
  - Teva Investigational Site 14200, Providence, Rhode Island
  - Teva Investigational Site 14300, Charleston, South Carolina
  - Teva Investigational Site 14196, Greenville, South Carolina
  - Teva Investigational Site 14188, San Antonio, Texas
  - Teva Investigational Site 14192, San Antonio, Texas
  - Teva Investigational Site 14189, San Antonio, Texas
  - Teva Investigational Site 14190, Greenfield, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the study protocol and the statistical analysis plan. Requests will be reviewed for scientific merit, product approval status, and conflicts of interest. Patient level data will be de-identified and study documents will be redacted to protect the privacy of trial participants and to protect commercially confidential information. Please email USMedInfo@tevapharm.com to make your request.

RESULTS

PARTICIPANT FLOW:
Groups:
- Concurrent Control (CC): Participants were treated with their standard of care albuterol-administering reliever inhalers and did not use the digital system during the treatment period. Participants were reimbursed or given a voucher to use to purchase their existing reliever medications.
- Digital System (DS): Participants were trained on the use of the albuterol multidose dry powder inhaler with integrated electronic module (eMDPI) DS (including instructions on how to use both the eMDPI and the Smart Device Application [App]) and, upon demonstrating competency, received 2 albuterol eMDPI devices for use as reliever bronchodilators to replace their reliever treatment during the study. The eMDPI DS consisted of 4 devices: Device 1: albuterol eMDPI (the test investigational medicinal product [IMP]); Device 2: Patient-facing App; Device 3: Digital health platform (DHP) (Cloud solution); and Device 4: Provider-facing Dashboard. Participants received 90 micrograms (mcg) albuterol, 1 to 2 oral inhalations every 4 to 6 hours, as needed for 12 weeks.
Period: Overall Study
Arm/Group | Concurrent Control (CC) | Digital System (DS)
Started (Intent-to-treat (ITT) analysis set: included all randomized participants) | 166 | 167
Safety Analysis Set (All participants in the DS group who receive at least 1 dose of IMP and all participants in the CC group.) | 166 | 150
Modified Intent-to-treat (mITT) Analysis Set (Al participants who received at least 1 dose of IMP and at least 1 postbaseline assessment on any of the study endpoints.) | 163 | 150
Completed | 162 | 149
Not Completed | 4 | 18
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Protocol deviation | 1 | 4
Not completed — Lost to Follow-up | 2 | 5
Not completed — Other than specified | 1 | 8

BASELINE CHARACTERISTICS:
Population: ITT analysis set included all randomized participants.
Groups:
- Digital System (DS): Participants were trained on the use of the albuterol eMDPI DS (including instructions on how to use both the eMDPI and the App) and, upon demonstrating competency, received 2 albuterol eMDPI devices for use as reliever bronchodilators to replace their reliever treatment during the study. The eMDPI DS consisted of 4 devices: Device 1: albuterol eMDPI (the test IMP); Device 2: Patient-facing App; Device 3: DHP (Cloud solution); and Device 4: Provider-facing Dashboard. Participants received 90 mcg albuterol, 1 to 2 oral inhalations every 4 to 6 hours, as needed for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Concurrent Control (CC) | Digital System (DS) | Total
Number analyzed (Participants) | 166 | 167 | 333
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (16.61) | 43.9 (16.63) | 43.7 (16.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 120 | 230
  Male | 56 | 47 | 103
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 40 | 36 | 76
  Not Hispanic or Latino | 121 | 126 | 247
  Unknown or Not Reported | 5 | 5 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 124 | 116 | 240
  Race: Black or African American | 30 | 43 | 73
  Race: Asian | 4 | 2 | 6
  Race: Native Hawaiian or other Pacific Islander | 1 | 0 | 1
  Race: Not Reported | 6 | 5 | 11
  Race: Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Meaningful Asthma Improvement at the End of 12-Week Treatment Period
Description: Meaningful asthma improvement was defined as an Asthma Control Test (ACT) score of at least 20 at the end of the 12-week treatment period or an increase of at least 3 units on the ACT score from baseline at the end of the 12-week treatment period. The ACT was a simple, participant-completed tool used to assess overall asthma control. The 5 items included in the ACT assess daytime and night-time asthma symptoms, use of reliever medication, and impact of asthma on daily functioning. Each item in the ACT was scored on a 5-point scale, with a summation of all items providing scores ranging from 5 to 25. The scores span the continuum of poor control of asthma (score of 5) to complete control of asthma (score of 25), with a cutoff score of 19 and below indicating participants with poorly controlled asthma.
Time Frame: Baseline to Week 12
Population: mITT analysis set included all randomized participants who received at least 1 dose of IMP (IMP is albuterol eMDPI for the DS group and standard-of-care albuterol-administering rescue medication for the CC group) and at least 1 postbaseline assessment on any of the study endpoints.
Measure: Number; unit: percentage of participants
Arm/Group | Concurrent Control (CC) | Digital System (DS)
Number analyzed (Participants) | 163 | 150
percentage of participants | 54.6 | 61.33
Statistical Analysis 1: Comparison: Concurrent Control (CC) vs Digital System (DS); The statistical model is a logistic regression model with treatment group as a fixed factor, pooled study sites as a random factor, and baseline ACT score as a covariate; Test type: Other; Odds Ratio (OR) = 1.33

2. Secondary Outcome: Number of Discussions Between Participant and Investigational Center Healthcare Professional (iHCP) Regarding Inhaler Technique or Adherence
Description: Number of participants who had discussions with iHCP regarding inhaler technique or adherence are reported.
Time Frame: Baseline up to Week 12
Population: mITT analysis set included all randomized participants who received at least 1 dose of IMP (IMP is albuterol eMDPI for the DS group and standard-of-care albuterol-administering rescue medication for the CC group) and at least 1 postbaseline assessment on any of the study endpoints. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Concurrent Control (CC) | Digital System (DS)
Number analyzed (Participants) | 162 | 147
Participants
  No discussion | 121 | 87
  1 discussion | 38 | 39
  2 discussions | 3 | 7
  3 discussions | 0 | 6
  4 discussions | 0 | 4
  5 discussions | 0 | 4

3. Secondary Outcome: Number of Decreased Doses of Inhaled Medication
Description: Number of participants who received decreased dose of inhaled medication during the 12-week treatment period are reported.
Time Frame: Baseline up to Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Concurrent Control (CC) | Digital System (DS)
Number analyzed (Participants) | 163 | 150
Participants
  No decreased doses | 163 | 149
  1 decreased dose | 0 | 1

4. Secondary Outcome: Number of Increased Doses of Inhaled Medication
Description: Number of participants who received increased dose of inhaled medication during the 12-week treatment period are reported.
Time Frame: Baseline up to Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Concurrent Control (CC) | Digital System (DS)
Number analyzed (Participants) | 162 | 147
Participants
  No increased doses | 157 | 143
  1 increased dose | 4 | 3
  2 increased doses | 1 | 1

5. Secondary Outcome: Number of Changes to Different Inhaled Medication
Description: Number of participants who received different inhaled medication during the 12-week treatment period are reported.
Time Frame: Baseline up to Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Concurrent Control (CC) | Digital System (DS)
Number analyzed (Participants) | 162 | 147
Participants
  No change to different inhaled medication | 159 | 143
  1 change to different inhaled medication | 2 | 3
  2 changes to different inhaled medication | 1 | 1

6. Secondary Outcome: Number of Additional Inhaled Medication
Description: Number of participants who received additional inhaled medication during the 12-week treatment period are reported.
Time Frame: Baseline up to Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Concurrent Control (CC) | Digital System (DS)
Number analyzed (Participants) | 162 | 147
Participants
  No additional inhaled medication | 161 | 145
  1 additional inhaled medication | 1 | 2

7. Secondary Outcome: Number of Addition of a Systemic Corticosteroid Medication for Asthma Therapy
Description: Number of participants who received additional systemic corticosteroid medication for asthma therapy during the 12-week treatment period are reported.
Time Frame: Baseline up to Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Concurrent Control (CC) | Digital System (DS)
Number analyzed (Participants) | 162 | 147
Participants
  No addition of a systemic corticosteroid medication for asthma therapy | 159 | 140
  1 addition of a systemic corticosteroid medication for asthma therapy | 2 | 6
  2 addition of a systemic corticosteroid medication for asthma therapy | 1 | 1

8. Secondary Outcome: Frequency of Intervention to Manage Comorbid Conditions Associated With Poor Asthma Control
Description: Number of participants with different frequency of intervention to manage comorbid conditions such as Gastroesophageal Reflux Disease (GERD) and Sinusitis are reported.
Time Frame: Baseline up to Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Concurrent Control (CC) | Digital System (DS)
Number analyzed (Participants) | 162 | 147
Participants
  No intervention to manage comorbid conditions | 158 | 137
  Interventions taken 1 time to manage comorbid conditions | 3 | 9
  Interventions taken 2 times to manage comorbid conditions | 1 | 1

9. Secondary Outcome: Change From Baseline in Mean Weekly Short-acting Beta2 Agonist (SABA) Usage at Week 12 for the DS Group
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | Digital System (DS)
Number analyzed (Participants) | 148
mcg | -36.18 (125.519)

10. Secondary Outcome: Change From Baseline in the Number of SABA-free Days at Week 12 for the DS Group
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Digital System (DS)
Number analyzed (Participants) | 148
days | 1.4 (2.36)

11. Secondary Outcome: System Usability Scale (SUS) Overall Score
Description: The SUS was used to explore device acceptability and usability for participants in the DS group. It covered a variety of aspects of system usability, such as the need for support, training, and complexity, and thus giving a global view of subjective assessments of usability. It was a 10-question tool (with five response options; from 1=strongly disagree to 5=strongly agree) that provided a composite measure, ranging from 0 to 100, of the overall usability of the system being studied. Higher scores represent better usability level for the tool.
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Digital System (DS)
Number analyzed (Participants) | 139
units on a scale | 79.8 (15.68)

12. Secondary Outcome: Change From Baseline in Beliefs About Medicines Questionnaire (BMQ) Concern Subscale Score at Week 12
Description: The BMQ was used to assess cognitive representations of medicine. The Beliefs About Medicines Questionnaire-Specific 11 (BMQ-S11) was an 11-item questionnaire that assessed the representation of medication prescribed for personal use and the BMQ-General assesses beliefs about medicines in general. BMQ concern is a 6-item scale assessing participant's concerns about potential adverse consequences (range: 1=strongly disagree to 5=strongly agree). Participants indicated their degree of agreement on a 5-point scale, ranging from 1=strongly disagree to 5=strongly agree. Scores obtained for individual items were summed, divided by the total number of items and multiplied by 5 to give a total score ranging from 5 to 25 (higher scores=stronger beliefs).
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Concurrent Control (CC) | Digital System (DS)
Number analyzed (Participants) | 153 | 135
units on a scale | -0.35 (3.767) | -0.72 (4.485)

13. Secondary Outcome: Change From Baseline in BMQ Necessity Subscale Score at Week 12
Description: The BMQ was used to assess cognitive representations of medicine. The Beliefs About Medicines Questionnaire-Specific 11 (BMQ-S11) was an 11-item questionnaire that assessed the representation of medication prescribed for personal use and the BMQ-General assesses beliefs about medicines in general. BMQ necessity is a 5-item scale assessing participant's beliefs about necessity of medications for controlling disease. Participants indicated degree of agreement on a 5-point scale, ranging from 1=strongly disagree to 5=strongly agree. Scores obtained for individual items were summed, divided by the total number of items and multiplied by 5 to give a total score ranging from 5 to 25 (higher scores=stronger beliefs).
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Concurrent Control (CC) | Digital System (DS)
Number analyzed (Participants) | 153 | 135
units on a scale | -0.2 (3.69) | -0.9 (3.99)

14. Secondary Outcome: Change From Baseline in Brief Illness Perception Questionnaire (BIPQ) Illness Comprehensibility Subscale Score at Week 12
Description: The BIPQ was a 9-item questionnaire designed to rapidly assess cognitive and emotional representations of illness. Only one item assesses illness comprehensibility or coherence of illness (Item 7: How well do you feel you understand your illness?). This item was rated using a 0 (do not understand at all) to 10 (understand very clearly) response scale. A higher score indicates a stronger illness comprehensibility.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Concurrent Control (CC) | Digital System (DS)
Number analyzed (Participants) | 153 | 135
units on a scale | 0.1 (2.30) | 0.2 (1.64)

15. Secondary Outcome: Change From Baseline in BIPQ Cognitive Subscale Score at Week 12
Description: BIPQ was a 9-item questionnaire designed to rapidly assess cognitive and emotional representations of illness. It comprised 5 items on cognitive representation of illness perception: consequences (Item 1: How much does your illness affect your life? Response range 0 [no affect] - 10 [severe affect]), timeline (Item 2: How long do you think your illness will continue? Response range 0 [a very short time] - 10 [forever]), personal control (Item 3: How much control do you feel you have over your illness? Response range 0 [no control] - 10 [extreme amount of control]), treatment control (Item 4: How much do you think your treatment can help your illness? Response range 0 [not at all] - 10 [extremely helpful]), and identity (Item 5: How much do you experience symptoms from your illness? Response range 0 [no symptoms] - 10 [severe symptoms]). Total BIPQ Cognitive Subscale Score was the sum of all item score and ranged from 0 to 50. A higher score indicates stronger illness perception.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Concurrent Control (CC) | Digital System (DS)
Number analyzed (Participants) | 153 | 135
units on a scale | -1.6 (5.32) | -2.0 (5.13)

16. Secondary Outcome: Change From Baseline in BIPQ Emotional Representations Subscale Score at Week 12
Description: BIPQ was a 9-item questionnaire designed to rapidly assess cognitive and emotional representations of illness. It comprised 2 items on emotional representation: concern (Item 6: How concerned are you about your illness? Response range 0 [not at all concerned] - 10 [extremely concerned]) and emotions (Item 8: How much does your illness affect you emotionally; for example, does it make you angry, scared, upset or depressed? Response range 0 [not at all affected emotionally] - 10 [extremely affected emotionally]). Total BIPQ Emotional Subscale Score was the sum of above 2 items score and ranged from 0 to 20. A higher score indicates extreme emotional representation.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Concurrent Control (CC) | Digital System (DS)
Number analyzed (Participants) | 153 | 135
units on a scale | -1.1 (3.76) | -0.8 (4.11)

17. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. SAEs included death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized the participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A summary of serious and non-serious AEs regardless of causality is located in 'Reported Adverse Events module'. Number of participants with any AEs, treatment-related AEs, and device-related AEs has been reported.
Time Frame: Baseline up to Week 14
Population: Safety analysis set included all participants in the DS group who received at least 1 dose of IMP and all participants in the CC group.
Measure: Count of Participants; unit: Participants
Arm/Group | Concurrent Control (CC) | Digital System (DS)
Number analyzed (Participants) | 166 | 150
Participants
  Any AEs | 26 | 28
  Treatment-related AE | 0 | 1
  Device-related AEs | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Week 14
Description: Safety analysis set included all participants in the DS group who received at least 1 dose of IMP and all participants in the CC group.
Arm/Group | Concurrent Control (CC) | Digital System (DS)
All-Cause Mortality (participants affected / at risk) | 0/166 | 0/150
Serious Adverse Events (participants affected / at risk) | 1/166 | 1/150
Other Adverse Events (participants affected / at risk) | 8/166 | 11/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Concurrent Control (CC) (N=166) | Digital System (DS) (N=150)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
SARS-CoV-2 sepsis (Infections and infestations) | 1 (1) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Concurrent Control (CC) (N=166) | Digital System (DS) (N=150)
Asthma (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 11 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2021-03-12): https://cdn.clinicaltrials.gov/large-docs/66/NCT03890666/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-13): https://cdn.clinicaltrials.gov/large-docs/66/NCT03890666/SAP_001.pdf